CLINICAL TRIAL: NCT03311763
Title: A Multi-center Exercise Intervention for Persons Transitioning to Dialysis Using the "Exercise is Medicine" Framework
Brief Title: Exercise is Medicine for Patients With CKD
Acronym: EIM-CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Emory University (Other); Santa Clara Valley Medical Center (Other)
Responsible Party: Principal Investigator, Shuchi Anand, Instructor in Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-43198
Record Dates: First submitted 2017-10-09; First posted 2017-10-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Disease stage4; Chronic Kidney Disease Stage V; Physical Activity
Keywords: implementation
MeSH Terms: conditions — Motor Activity | interventions — Counseling; Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Counseling alone (Active Comparator): Group 1: physical activity assessment, brief counseling session + physical activity wearable
  Interventions: Behavioral: Counseling and wearable device
- Group exercise (Experimental): Group 2: Group 1 intervention components + referral to a free, community-based, EIM practitioner led group exercise program (two, 1 hour classes/week for 8 weeks).
  Interventions: Behavioral: EIM Fitness Practitioners; Behavioral: Counseling and wearable device

INTERVENTIONS:
Behavioral: EIM Fitness Practitioners — Exercise is Medicine Practitioners will facilitate peer groups that attend twice-weekly exercise classes for 8 weeks, with clinical monitoring and advise regarding increasing physical activity.
  Arms: Group exercise
Behavioral: Counseling and wearable device — Brief exercise counseling session and provision of a wearable fitness tracking device to promote physical activity.

SUMMARY:
The investigators plan to integrate and tailor the existing Exercise is Medicine framework, an evidence-based multi-level intervention program developed by the American Society of Sports Medicine, for the care of patients with advanced chronic kidney disease. In this pilot randomized control trial, investigators will compare the effects and feasibility of two intervention arms designed to start and maintain physical activity in this high-risk population (Group 1: physical activity assessment, brief counseling session + physical activity wearable versus Group 2: Group 1 intervention components + referral to a free, community-based, EIM practitioner led group exercise program).

DETAILED DESCRIPTION:
Persons on dialysis are physically inactive, with most reporting activity levels below the fifth percentile of healthy age-matched groups. Physical inactivity in turn increases the risk for functional decline and mortality in this vulnerable population. The investigators propose a pragmatic clinical trial for an exercise intervention among persons transitioning to dialysis. The investigators will use an existing framework - Exercise is Medicine (EIM) - developed by the American College of Sports Medicine. The investigators will randomize 98 persons from two regions-Atlanta and Bay Area-in two intervention arms with incremental levels of clinical-community integration: physical activity assessment during Nephrology clinical visit, brief counseling at pre-dialysis education and physical activity wearable (group 1) versus group 1 intervention components plus a referral to a free, EIM practitioner-led group exercise program over 16 weeks (group 2; 8 week core intervention; 8 week follow up). The investigators will assess efficacy by comparing between group differences in minutes/week of (measured) moderate intensity physical activity. To evaluate implementation, investigators will use questionnaires and exit interviews for assessing barriers to referral, participation and retention along the path of the intervention; investigators will use cost-utility analyses to assess scalability. Further the investigators will have a plan for dissemination of the intervention by partnering with insurance providers and both for-profit and non-profit dialysis organizations. The overall goal is to inform the development of a practical, cost-conscious intervention that addresses barriers to physical activity commonly faced by persons on dialysis, and can be delivered as a "package" to interested practices.

ELIGIBILITY:
Inclusion Criteria:

* - eGFR < 30 ml/min/1.73m2
* Age ≥30 and ≤80 years
* Noncompliance with physical activity guidelines
* Not in precontemplation stage
* Non-wheelchair bound
* Able to provide informed consent in English or Spanish
* Anticipated to be living in the area over the next 36 weeks

Exclusion Criteria:

* - Inability to provide consent in English
* Diagnosed mental health disorder
* Alcohol or drug abuse
* No fixed address or contact details
* Unstable angina or unstable arrhythmias
* Lack of access to internet
* Any concern not otherwise stated by patient's nephrologist

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Differences in minutes of physical activity per week as measured by wearable device | measured at baseline, 8 weeks and 16 weeks post start of intervention.
  The Garmin wearable device will be used to track physical activity minutes during the week, with differences in total minutes per week in baseline versus 8 weeks (and 16 weeks) post intervention compared between exercise classes versus counseling alone groups

SECONDARY OUTCOMES:
Six minute walk test (6MWT) | measured at baseline, 8 weeks and 16 weeks post start of intervention.
  6 minute walk test will be administered by research personnel in 100 feet walkway, with differences in distance walked between baseline and 8 weeks (and 16 weeks), compared between group exercise and counseling alone groups
Handgrip | measured at baseline, 8 weeks and 16 weeks post start of intervention.
  Dynamometers will be used to measure handgrip strength, with differences in distance walked between baseline and 8 weeks (and 16 weeks), compared between group exercise and counseling alone groups
Health-related Quality of life using Medical Outcomes Short form 12 | measured at baseline, 8 weeks and 16 weeks post start of intervention.
  Questionnaire based Sf12 will be used to measure health related quality of life, with differences in distance walked between baseline and 8 weeks (and 16 weeks), compared between group exercise and counseling alone groups

OTHER OUTCOMES:
Symptoms of Depression as measured by Center for Epidemiologic Studies Depression Scale (CESD20) | measured at baseline, 8 weeks and 16 weeks post start of intervention.
  Questionnaire based CESD-2 scale will be used to measure depression
Physical activity self-efficacy questionnaire | measured at baseline, 8 weeks and 16 weeks post start of intervention.
Waist circumference | measured at baseline, 8 weeks and 16 weeks post start of intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Clara Valley Nephrology, San Jose, California
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anand S, Ziolkowski SL, Bootwala A, Li J, Pham N, Cobb J, Lobelo F. Group-Based Exercise in CKD Stage 3b to 4: A Randomized Clinical Trial. Kidney Med. 2021 Jul 8;3(6):951-961.e1. doi: 10.1016/j.xkme.2021.04.022. eCollection 2021 Nov-Dec. PMID 34939004
- [Background] Jagannathan R, Ziolkowski SL, Weber MB, Cobb J, Pham N, Long J, Anand S, Lobelo F. Physical activity promotion for patients transitioning to dialysis using the "Exercise is Medicine" framework: a multi-center randomized pragmatic trial (EIM-CKD trial) protocol. BMC Nephrol. 2018 Sep 12;19(1):230. doi: 10.1186/s12882-018-1032-0. PMID 30208854